CLINICAL TRIAL: NCT00685139
Title: A Relative Bioavailability Study of 100 mg Zonisamide Capsules Under Fasting Conditions
Brief Title: Fasting Bioavailability Study of Zonisamide Capsules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Kristin Arnold, Vice President R&D, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: R04-1376
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Results first posted 2009-12-30 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Therapeutic Equivalency
MeSH Terms: interventions — Zonisamide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zonisamide 100 mg Capsule (Experimental): A single dose of zonisamide 100 mg administered after an overnight fast.
  Interventions: Drug: Zonisamide 100 mg Capsule
- Zonisamide (Zonegran® ) 100 mg Capsule (Experimental): A single dose of Zonegran® 100 mg administered after an overnight fast.
  Interventions: Drug: Zonisamide (Zonegran®) 100 mg Capsule

INTERVENTIONS:
Drug: Zonisamide 100 mg Capsule — 100 mg capsule administered after an overnight fast.
  Arms: Zonisamide 100 mg Capsule
Drug: Zonisamide (Zonegran®) 100 mg Capsule — 100 mg capsule administered after an overnight fast.
  Other Names: Zonegran®
  Arms: Zonisamide (Zonegran® ) 100 mg Capsule

SUMMARY:
The purpose of this study is to evaluate and compare the relative bioavailability of a test formulation of zonisamide capsules to an equivalent dose of a reference formulation, Zonegran® (zonisamide) capsules, after a single oral dose administered under fasting conditions.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate and compare the relative bioavailability of a test formulation of zonisamide capsules to an equivalent dose of a reference formulation, Zonegran® (zonisamide) capsules, after a single oral dose administered under fasting conditions.

Thirty-four healthy, non-smoking, non-obese male and female volunteers at least 18 years of age will be randomly assigned in a crossover fashion to receive each of two zonisamide dosing regimens in sequence with a 28 day washout period between dosing periods. On the morning of Day 1, after an overnight fast, subjects will receive either a single oral dose of the test formulation, zonisamide (1 x 100 mg capsule) or a single oral dose of the reference formulation, Zonegran® (1 x 100 mg capsule). After a 28 day washout period, on the morning of Day 29 after an overnight fast, subjects will receive the alternate regimen. Blood samples will be drawn from all participants before dosing and for 72 hours post dose at times sufficient to adequately define the pharmacokinetics of zonisamide. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout the confinement portion of the study for adverse reactions to the study drug and/or procedures. Blood pressure and heart rate will be obtained prior to dosing and as scheduled following dose administration. All adverse events whether elicited by query, spontaneously reported or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics:
* All volunteers selected for this study will be healthy men and women 18 years of age or older at the time of dosing
* Weight range will not exceed ± 20% for height and body frame
* Screening Procedures:
* Each volunteer will complete the screening process within 28 days prior to Period I dosing
* Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures
* Screening will include general observation, physical examination, demographics, medical and medication history, an electrocardiogram, sitting blood pressure and heart rate, respiratory rate and temperature
* The physical examination will include, but may not be limited to, an evaluation of the cardiovascular, gastrointestinal, respiratory and central nervous systems
* The screening clinical laboratory procedures will include: Hematology, Clinical Chemistry, HIV antibody, Hepatitis B-surface antigen, Hepatitis C antibody, Urinalysis, Urine Drug Screen, Serum Pregnancy Screen, Follicle Stimulating Hormone
* If female: postmenopausal for 1 year or surgically sterile.

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant
* Volunteers demonstrating a reactive screen for hepatitis B surface antigen, hepatitis C antibody or HIV antibody screen
* Volunteers demonstrating a positive drug abuse screen when screened for this study
* Female volunteers demonstrating a positive pregnancy screen
* Female volunteers who are currently breastfeeding
* Volunteers with a history of allergic response(s) to zonisamide or related drugs
* Volunteers with a history of clinically significant allergies including drug allergies
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigator)
* Volunteers who currently use tobacco products
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing
* Volunteers who report donating greater than 150mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for four weeks after completing the study
* Volunteers who report receiving any investigational drug within 14 days prior to Period I dosing.
* Volunteers who have donated plasma(e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for four weeks after completing the study
* Volunteers who report taking any systemic prescription medication in the 14 days prior to Period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-01; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Zonisamide 100 mg Capsules Then Zonegran® 100 mg Capsules: On the morning of Day 1 subjects received one capsule of the test formulation, zonisamide 100 mg, after an overnight fast, followed by a 28 day washout period. On the morning of Day 29 subjects received one capsule of the reference formulation, Zonegran® 100 mg, after an overnight fast.
- Zonegran® 100 mg Capsules Then Zonisamide 100 mg Capsules: On the morning of Day 1 subjects received one capsule of the reference formulation, Zonegran® 100 mg, after an overnight fast, followed by a 28 day washout period. On the morning of Day 29 subjects received one capsule of the test formulation, zonisamide 100 mg, after an overnight fast.
Period: First Intervention
Arm/Group | Zonisamide 100 mg Capsules Then Zonegran® 100 mg Capsules | Zonegran® 100 mg Capsules Then Zonisamide 100 mg Capsules
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0
Period: Washout Period of 28 Days
Arm/Group | Zonisamide 100 mg Capsules Then Zonegran® 100 mg Capsules | Zonegran® 100 mg Capsules Then Zonisamide 100 mg Capsules
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Zonisamide 100 mg Capsules Then Zonegran® 100 mg Capsules | Zonegran® 100 mg Capsules Then Zonisamide 100 mg Capsules
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Zonisamide 100 mg Capsules and Zonegran® 100 mg Capsules: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 29, each subject received one capsule of either zonisamide 100 mg or Zonegran® 100 mg following an overnight fast.
Arm/Group | Zonisamide 100 mg Capsules and Zonegran® 100 mg Capsules
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 33.6 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 31
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that the drug reaches in the plasma.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to dose administration (0 hour) and at 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5, 5, 5.5, 6, 6.5, 7, 8, 10, 12, 16, 24, 36, 48, 60 and 72 hours after drug administration.
Population: Pharmacokinetic analyses are based on 33 out of 34 subjects who completed this study. One subject elected to withdraw prior to the study hour 2 blood sample collection during period II.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Zonisamide 100 mg Capsules; Zonegran® 100 mg Capsules: On the morning of Day 1 subjects received one capsule of the test formulation, zonisamide 100 mg, or the reference formulation, Zonegran® 100 mg, after an overnight fast followed by a 28 day washout period. On the morning of Day 29 subjects received the alternate regimen following an overnight fast.
Arm/Group | Zonisamide 100 mg Capsules | Zonegran® 100 mg Capsules
Number analyzed (Participants) | 33 | 33
ng/mL | 1,052.65 (348.13) | 1,078.46 (417.66)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Zonisamide 100 mg Capsules | Zonegran® 100 mg Capsules
Number analyzed (Participants) | 33 | 33
ng-hr/mL | 42,338.31 (11,202.96) | 42,873.95 (11,964.12)

ADVERSE EVENTS:
Groups:
- Zonisamide 100 mg Capsules: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 29, each subject received one capsule of either zonisamide 100 mg or Zonegran 100 mg following an overnight fast.
- Zonegran® 100 mg Capsules: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 29, each subject received one capsule of either zonisamide 100 mg or Zonegran® 100 mg following an overnight fast.
Arm/Group | Zonisamide 100 mg Capsules | Zonegran® 100 mg Capsules
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 5/34 | 3/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide 100 mg Capsules (N=34) | Zonegran® 100 mg Capsules (N=34)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Haematoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days